CLINICAL TRIAL: NCT01154881
Title: A Trial Evaluating the Pharmacodynamic Response of NN1250 at Steady State in Subjects With Type 2 Diabetes
Brief Title: A Trial Evaluating the Blood Glucose-lowering Effect of NN1250 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-1987; U1111-1114-9099 (Other: WHO); 2009-017281-23 (EudraCT Number)
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- IDeg 100U/mL 0.4U/kg (Experimental)
  Interventions: Drug: insulin degludec
- IDeg 100U/mL 0.6U/kg (Experimental)
  Interventions: Drug: insulin degludec
- IDeg 100U/mL 0.8U/kg (Experimental)
  Interventions: Drug: insulin degludec
- IDeg 200U/mL 0.6U/kg (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Insulin degludec (IDeg) injected s.c. (under the skin) once daily for 6 days in each treatment period. Each subject was randomly allocated to 2 out of 4 treatments.

SUMMARY:
This trial was conducted in Europe. The aim of this clinical trial was to evaluate the blood glucose-lowering effect of NN1250 (insulin degludec/insulin 454) in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index (BMI) below or equal to 35.0 kg/m2

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve from 0-24 hours at steady state | 0-24 hours (derived on treatment day 6)

SECONDARY OUTCOMES:
Area under the insulin degludec concentration-time curve from 0-24 hours at steady state | 0-24 hours (derived on treatment day 6)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Nosek L, Bottcher SG, Hastrup H, Haahr H. Ultra-long-acting insulin degludec has a flat and stable glucose-lowering effect in type 2 diabetes. Diabetes Obes Metab. 2012 Oct;14(10):944-50. doi: 10.1111/j.1463-1326.2012.01638.x. Epub 2012 Jul 10. PMID 22726241
- [Result] Heise T, Korsatko S, Nosek L, Coester HV, Deller S, Roepstorff C, Segel S, Kapur R, Haahr H, Hompesch M. Steady state is reached within 2-3 days of once-daily administration of degludec, a basal insulin with an ultralong duration of action. J Diabetes. 2016 Jan;8(1):132-8. doi: 10.1111/1753-0407.12266. Epub 2015 Mar 24. PMID 25581159
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com